CLINICAL TRIAL: NCT03636789
Title: Evaluation of the Prevalence of Oculomotor Disorders in Patients With Radiologically Isolated Syndrome
Acronym: OCRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2017-01/GC-01
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Radiologically Isolated Syndrome (RIS); Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurological consultation group (Experimental)
  Interventions: Other: Neurological consultation

INTERVENTIONS:
Other: Neurological consultation — study of horizontal, vertical, reflex and voluntary saccades, and of horizontal and vertical ocular pursuit by a BrainTracker eye-oculography system

SUMMARY:
This study aims to investigate the prevalence of subclinical oculomotor disorders in a population of patients with radiologically isolated syndrome.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his informed consent and signed the consent form.
* The patient must be affiliated or beneficiary of a health insurance plan.
* The patient is at least 18 years old (≥) and under 50 years old (≤).
* Patients with radiologically isolated syndrome according to the criteria of Okuda et al. (2009)
* Diagnosis of a radiologically isolated syndrome confirmed by the national expert center of Nice for less than 3 years.

Exclusion Criteria:

* The subject participates in another study.
* The subject is in an exclusion period determined by a previous study.
* The subject is under guardianship, curatorship or safeguard of justice.
* The patient is pregnant or breastfeeding
* The subject refuses to sign the consent.
* It is not possible to give the subject informed information.
* Patient presenting a pathological neurological examination.
* Patient with visual acuity less than 5/10 or with ocular instability

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the occurrence of oculomotor disorders | Day 0
  using a video-oculographic recording system

SECONDARY OUTCOMES:
To establish the prevalence of each of the different types of oculomotor abnormalities that constitute the oculomotor disorder | Day 0
  number
To identify a correlation between oculomotor disorders and MRI abnormalities. | Day 0
To identify a correlation between oculomotor disorders and the cognitive impairment test (Symbol Digit Modalities Test) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Castelnovo, Principal Investigator — Nîmes University Hospital
Locations (6):
- France (6):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Hôpital Guy de Chauliac, Montpellier
  - Nice University Hospital, Nice
  - Nimes University Hospital, Nîmes
  - Pitié Salpêtrière University Hospital (APHP), Paris
  - Toulouse University Hospital, Toulouse